CLINICAL TRIAL: NCT01768871
Title: Prospective, Long-Term, Multi-Center Study on the Efficacy of the VEGA System® for Total Knee Arthroplasty.
Brief Title: Evaluation of the VEGA Knee System® Range of Motion
Status: Terminated | Type: Observational
Why Stopped: low enrollment
Sponsor: Aesculap Implant Systems (Industry)
Responsible Party: Sponsor
Other Study IDs: AAG-O-H-1105
Record Dates: First submitted 2013-01-14; First posted 2013-01-16 (Estimated); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Patients With Total Knee Arthroplasty Using the VEGA System

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary objective of this study is to evaluate the function of the knee after a total knee replacement with the VEGA system®.

DETAILED DESCRIPTION:
To evaluate patients after total knee arthroplasty in terms of function for five years.

ELIGIBILITY:
Inclusion Criteria:

* willing to sign the informed consent.
* Patient has intact collateral ligaments.

Exclusion Criteria:

* Inflammatory arthritis
* Patients that have had a high tibial osteotomy or femoral osteotomy
* Patients with neuromuscular or neurosensory deficiency which would make it difficult to assess the device performance.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have undergone a total knee arthroplasty with the VEGA knee system®
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2013-01; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
WOMAC | Two years
  WOMAC function score 2 years post arthroplasty

SECONDARY OUTCOMES:
Health related quality of life | Two years

CONTACTS AND LOCATIONS:
Overall Officials: Khaled Saleh, Study Chair — Southern Illinois University School of Medicine
Locations (3):
- United States (3):
  - Rose Medical Center, Denver, Colorado
  - DBA Hussamy Sports and Hand Center, Vero Beach, Florida
  - Charles J DePaolo, MD, PA, Asheville, North Carolina